CLINICAL TRIAL: NCT02038569
Title: Effect of Calcipotriol Plus Betamethasone Dipropionate Gel on the HPA Axis and Calcium Metabolism in Adolescent Subjects (Aged 12 to 16 Years, 11 Months) With Scalp and Body Psoriasis
Brief Title: An International, Multi-centre, Prospective, Non-controlled, Open, Single-group, 8-week Trial in Adolescent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0076-1017
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 80185 gel (Experimental)
  Interventions: Drug: LEO 80185 gel

INTERVENTIONS:
Drug: LEO 80185 gel

SUMMARY:
An international, multi-centre, prospective, non-controlled, open, single-group, 8-week trial in adolescent subjects (aged 12 to 16 years, 11 months) with scalp and body psoriasis.

DETAILED DESCRIPTION:
A phase 2 trial evaluating the safety and efficacy of once daily use of LEO 80185 gel containing calcipotriol 50 mcg/g plus betamethasone 0.5mg/g (as dipropionate) in adolescent subjects (aged 12 to 16 years, 11 months) with scalp and body psoriasis.

ELIGIBILITY:
Inclusion Criteria (all subjects):

* Clinical signs of psoriasis vulgaris on both the scalp and body (trunk and/or limbs)
* At SV2 and Visit 1, a clinical diagnosis of scalp and body (trunk and/or limbs) psoriasis which is:

  * of an extent of 10 to 35% of the body surface area (excluding psoriatic lesions of the face and sensitive areas. Sensitive areas include armpits, groin, under the breasts and in other skin folds around the genitals and buttocks), and
  * of at least moderate severity according to the investigator's global assessment of disease severity on the body.
* A serum albumin-corrected calcium level below the upper reference limit at SV2

Inclusion Criteria (for subjects performing HPA axis assessments):

* At SV2 and Visit 1, a clinical diagnosis of scalp psoriasis which is:

  * more than or equal to 20% of the scalp area, and
  * of at least moderate severity according to the investigator's global assessment of disease severity on the scalp.
* Subjects with a normal HPA axis function at SV2 including serum cortisol concentration above 5 mcg/dl before ACTH challenge and serum cortisol concentration above 18 mcg/dl 30 minutes after ACTH challenge.

Inclusion Criteria (for subjects not performing HPA axis assessments):

* At SV2 and Visit 1, a clinical diagnosis of scalp psoriasis which is:

  * more than or equal to 10% of the scalp area, and
  * of at least moderate severity according to the investigator's global assessment of disease severity on the scalp.

Exclusion Criteria (all subjects):

* Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on scalp and/or body psoriasis within the following time period prior to Visit 1 and during the trial:

  * etanercept - within 4 weeks prior to Visit 1
  * adalimumab, infliximab - within 2 months prior to Visit 1
  * ustekinumab - within 4 months prior to Visit 1
  * experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to Visit 1
* Systemic treatment with therapies other than biologicals, with a possible effect on scalp and/or body psoriasis (e.g., retinoids, immunosuppressants, PUVA) within 4 weeks prior to Visit 1 (Day 0) or during the trial.
* UVB therapy within 2 weeks prior to Visit 1 or during the trial.
* Any topical treatment on the scalp and body (except for emollients and non-steroid medicated shampoos) within 2 weeks prior to Visit 1 or during the trial.
* Systemic calcium, vitamin D supplements, antacids, diuretics, antiepileptics, diphosphonates or calcitonin within 4 weeks prior to SV2 or during the trial.
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis (e.g., betablockers, chloroquine, lithium, ACE inhibitors) during the trial.
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
* Subjects with any of the following conditions present on the treatment areas on scalp and/or body: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds.
* Other inflammatory skin diseases that may confound the evaluation of scalp and/or body psoriasis.
* Planned excessive exposure to sun during the trial that may affect scalp and/or body psoriasis.
* Known or suspected severe renal insufficiency or severe hepatic disorders.
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia.
* Any clinically significant abnormality following review of screening laboratory tests (blood and urine samples), physical examination or blood pressure/heart rate measurement performed at SV2.
* Current participation in any other interventional clinical trial.
* Previously enrolled in this trial.
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within a month prior to SV1 or longer, if the class of substance required a longer wash-out as defined above (e.g., biological treatments).
* Subjects or parent(s) or legal guardian known or suspected of being unlikely to comply with the Clinical Trial Protocol (e.g., alcoholism, drug dependency or psychotic state).
* Females who are pregnant, or of child-bearing potential and wishing to become pregnant during the trial, or who are breast-feeding.
* Females of child-bearing potential with positive pregnancy test at SV2.
* Subject (or their partner) not using an adequate method of contraception according to national requirements.

Exclusion Criteria (for subjects performing HPA axis assessments)

* A history of serious allergy, allergic asthma or serious allergic skin rash.
* Known or suspected hypersensitivity to any component of CORTROSYN® (including ACTH/cosyntropin/tetracosactide)
* Systemic treatment with corticosteroids (including inhaled and nasal steroids) within 12 weeks prior to SV2 or during the trial.
* Topical treatment with corticosteroids within 2 weeks prior to SV2 or during the trial.
* Oestrogen therapy (including contraceptives) or any other medication known to affect cortisol levels levels or HPA axis integrity within 4 weeks prior to SV2 or during the trial.
* Enzymatic inductors (e.g., barbiturates, phenytoin, rifampicin) within 4 weeks prior to SV2 or during the trial.
* Systemic or topical cytochrome P450 inhibitors (e.g., ketoconazole, itraconazole, metronidazole) within 4 weeks prior to SV2 or during the trial. Topical ketoconazole 2 weeks prior to SV2.
* Hypoglycemic sulfonamides within 4 weeks prior to SV2 or during the trial.
* Antidepressive medications within 4 weeks prior to SV2 or during the trial.
* Known or suspected endocrine disorder that may affect the results of the ACTH challenge test.
* Clinical signs or symptoms of Cushing's disease or Addison's disease.
* Subjects with diabetes mellitus.
* Known or suspected cardiac condition.
* Not following nocturnal sleep patterns.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Eichenfield, MD, Principal Investigator — Rady Chilidren's Hospital
Locations (35):
- United States (8):
  - Rady's Children Hospital, San Diego, California
  - Clinical Research Center, Morsani Center for Advanced Healthcare, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Skin Specialists, PC, Omaha, Nebraska
  - St. Luke's Roosevelt Hospital, Forest Hills, New York
  - Clinical Partners, Johnston, Rhode Island
  - Dermatology and Laser Center of Charleston, PA, Charleston, South Carolina
  - Clinical Trials of Texas, Inc., San Antonio, Texas
- Canada (4):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Adult, Pediatric and Laser Derma, St. John's, Newfoundland and Labrador
  - Lynderm Research Inc., Markham, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
- France (3):
  - CHU de Nice, Nice, Alpe-Maritimes
  - Cabinet Medical, Martigues, Bouches-du-Rhône
  - CHI de Cornouaille, Quimper, Finistère
- Germany (4):
  - Charite Berlin, Berlin
  - Uniklinik Bonn, Bonn
  - Uniklinik Frankfurt, Frankfurt am Main
  - Katholisches Kinderkrankenhaus, Hamburg
- Poland (5):
  - Endo - Med. Centrum Medyczne Clinic, Karczew
  - NZOZ Med.-Laser Clinic, Lublin
  - Specjalistyczny Ofrodek Leczniczo Clinic, Ostróda
  - Medycyna Kliniczna Clinic, Warsaw
  - Derm Medica Sp.zo.o. Clinic, Wroclaw
- Romania (7):
  - Policlinica de Diagnostic Rapid S.A. Clinic, Brasov
  - Spitalul Clinic "Colentina", Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Cabinet Medical Individual Tatu G. Alin Laurentiu, Galati
  - Iasiprest SRL Dermato-Venerology, Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- United Kingdom (4):
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Monklands Hospital, Airdrie, Lanarkshire
  - Whipps Cross University Hospital, Leytonstone, London
  - St. Woolos Hospital, Stow Hill, Newport, Monmouthshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LEO 80185 Gel: LEO 80185 gel, containing calcipotriol (50 mcg/g) and betamethasone (0.5 mg/g, as dipropionate), was applied once daily to scalp and body psoriasis lesions.
Period: Overall Study
Arm/Group | LEO 80185 Gel
Started | 107
Completed | 102
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- LEO 80185 Gel: LEO 80185 gel, containing calcipotriol (50 mcg/g) and betamethasone (0.5 mg/g, as dipropionate), was applied once daily to scalp and body psoriasis lesions. This arm contains all 107 subjects that were assigned to treatment and constitutes the full analysis set and the safety analysis set. 31 subjects in this arm performed additional hypothalamic-pituitary axis assessments and constitute the per protocol analysis set.
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 97
  Black or African American | 2
  Other | 2
  Asian | 6
Region of Enrollment [Number; unit: participants]
  Canada | 6
  Romania | 42
  United States | 12
  Poland | 14
  United Kingdom | 8
  France | 5
  Germany | 20
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is based on skin reaction to first 30-45 minutes sun exposure after a winter with no sun exposure:
  Type I: Unexposed skin color: white, always burns easily, never tans. Type II: Unexposed skin color: white, always burns easily, tans minimally. Type III: Unexposed skin color: white, burns moderately, tans gradually (light brown).
  Type IV: Unexposed skin color: white, burns minimally, always tans well (moderate brown).
  Type V: Unexposed skin color: brown, rarely burns, tans profusely (dark brown). Type VI: Unexposed skin color: black, never burns, deeply pigmented.
  Participants
    Type I | 2
    Type II | 47
    Type III | 34
    Type IV | 20
    Type V | 2
    Type VI | 2
Duration of psoriasis vulgaris [Mean (Standard Deviation); unit: years] | 4.1 (3.2)
Investigator's global assessment of disease severity on body [Count of Participants; unit: Participants]
  Mild | 14
  Moderate | 87
  Severe | 6
Psoriasis Area and Severity Index Score [Mean (Standard Deviation); unit: score on a scale] — Psoriasis area and severity index (PASI) assesses extent and severity of clinical signs of psoriasis vulgaris. Body surface is divided in 4 ares: head (incl. neck), arms (incl. hands), trunk (incl. flexures) and legs (incl. buttocks and feet). Each area is scored from 0-6 for extent of psoriasis and from 0-4 for redness, thickness, and scaliness, and an area PASI score is calculated. The total PASI score is calculated from each area's score. The PASI score ranges from 0 (clear skin) to 72 (maximum disease), a PASI score higher than 10 generally corresponds to moderate-to-severe disease.
  score on a scale | 10.70 (4.41)
Investigator's assessment of extent of psoriasis on the body and scalp (%) [Mean (Standard Deviation); unit: % of body surface area affected] | 14.9 (8.3)
Patient's global assessment of disease severity on body [Count of Participants; unit: Participants]
  Very Mild | 5
  Mild | 21
  Moderate | 77
  Severe | 4

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Reactions (ADRs)
Description: Number of Adverse Drug Reactions (ADRs)
Time Frame: 8 weeks
Population: Safety analysis set
Measure: Number; unit: Number of adverse drug reactions
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Number of adverse drug reactions
  Blood cortisol decreased | 2
  Blood parathyroid hormone increased | 1
  Acne | 1
  Erythema | 1
  Hyperparathyroidism | 1
  Folliculitis | 1
  Headache | 1

2. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After ACTH-challenge at Week 4
Description: Number of subjects with serum cortisol concentration of ≤18 mcg/dl at 30 minutes after ACTH-challenge at Week 4
Time Frame: 30 minutes after ACTH-challenge at Week 4
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Participants
  Serum cortisol equal to or below 18 mcg/dL | 4
  Serum cortisol above 18 mcg/dL | 27

3. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After ACTH-challenge at Week 8
Description: Number of subjects with serum cortisol concentration of ≤18 mcg/dl at 30 minutes after ACTH-challenge at Week 8
Time Frame: 30 minutes after ACTH-challenge at Week 8
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Participants
  Serum cortisol equal to or below 18 mcg/dL | 2
  Serum cortisol above 18 mcg/dL | 27
  No assessment performed | 2

4. Primary Outcome: Change in Albumin-corrected Serum Calcium From Baseline to Week 4
Description: Change in albumin-corrected serum calcium from baseline to Week 4
Time Frame: From baseline to Week 4
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/L | -0.012 (0.131)

5. Primary Outcome: Change in Albumin-corrected Serum Calcium From Baseline to Week 8
Description: Change in albumin-corrected serum calcium from baseline to Week 8
Time Frame: From baseline to Week 8
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/L | -0.008 (0.125)

6. Primary Outcome: Change in Albumin-corrected Serum Calcium From Baseline to End of Treatment
Description: Change in albumin-corrected serum calcium from baseline to end of treatment, defined as the last value recorded after baseline up to and including Week 8.
Time Frame: From baseline to end of treatment
Population: Safety analysis set.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/L | -0.003 (0.121)

7. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to Week 4
Description: Change in 24-hour urinary calcium excretion from baseline to Week 4
Time Frame: From baseline to Week 4
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/24hr | -0.493 (1.669)

8. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to Week 8
Description: Change in 24-hour urinary calcium excretion from baseline to Week 8
Time Frame: From baseline to Week 8
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/24hr | 0.040 (1.638)

9. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to End of Treatment
Description: Change in 24-hour urinary calcium excretion from baseline to end of treatment, defined as the last value recorded after baseline up to and including Week 8.
Time Frame: From baseline to end of treatment
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/24hr | 0.069 (1.593)

10. Secondary Outcome: Adverse Events (AEs)
Description: Number of Adverse Events (AEs)
Time Frame: 8 weeks
Population: Safety analysis set
Measure: Number; unit: Adverse Events
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Adverse Events
  Nasopharyngitis | 6
  Rhinitis | 2
  Folliculitis | 1
  Hordeolum | 1
  Impetigo | 1
  Peritonsillar abscess | 1
  Upper respiratory tract infection | 1
  Viral infection | 1
  Blood parathyroid hormone increased | 5
  Blood cortisol decreased | 2
  Eosinophil count increased | 1
  Headache | 8
  Balance disorder | 1
  Dizziness | 1
  Syncope | 1
  Cough | 2
  Oropharyngeal pain | 2
  Dyspnoea | 1
  Epistaxis | 1
  Respiratory disorder | 1
  Acne | 1
  Erythema | 1
  Pruritus | 1
  Sunburn | 1
  Abdominal pain upper | 1
  Constipation | 1
  Diarrhoea | 1
  Back pain | 1
  Muscle spasms | 1
  Musculoskeletal chest pain | 1
  Neck pain | 1
  Dysmenorrhoea | 3
  Arthropod sting | 1
  Concussion | 1
  Sleep disorder | 1
  Suicide attempt | 1
  Cardiovascular disorder | 1
  Hyperparathyroidism | 1
  Iron deficiency | 1
  Wisdom teeth removal | 1

11. Secondary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at Both 30 and 60 Minutes After ACTH-challenge at Week 4
Description: Number of subjects with serum cortisol concentration of ≤18 mcg/dl at both 30 and 60 minutes after ACTH-challenge at Week 4
Time Frame: 30 and 60 minutes after ACTH-challenge at Week 4
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Participants
  Serum cortisol equal to or below 18 mcg/dL | 0
  Serum cortisol above 18 mcg/dL | 31

12. Secondary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at Both 30 and 60 Minutes After ACTH-challenge at Week 8
Description: Number of subjects with serum cortisol concentration of ≤18 mcg/dl at both 30 and 60 minutes after ACTH-challenge at Week 8
Time Frame: 30 and 60 minutes after ACTH-challenge at Week 8
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Participants
  Serum cortisol equal to or below 18 mcg/dL | 0
  Serum cortisol above 18 mcg/dL | 29
  No assessment performed | 2

13. Secondary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to Week 4
Description: Change in urinary calcium:creatinine ratio from baseline to Week 4
Time Frame: From baseline to Week 4
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/g | -0.098 (1.642)

14. Secondary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to Week 8
Description: Change in urinary calcium:creatinine ratio from baseline to Week 8
Time Frame: From baseline to Week 8
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/g | 0.219 (1.700)

15. Secondary Outcome: Change in Serum Alkaline Phosphatase From Baseline to Week 4
Description: Change in serum alkaline phosphatase from baseline to Week 4
Time Frame: From baseline to Week 4
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/L | -0.4 (31.4)

16. Secondary Outcome: Change in Serum Alkaline Phosphatase From Baseline to Week 8
Description: Change in serum alkaline phosphatase from baseline to Week 8
Time Frame: From baseline to Week 8
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
mmol/L | -6.8 (42.6)

17. Secondary Outcome: Pharmacokinetic Evaluation AUC(0-t)
Description: AUC(0-t) values for betamethasone dipropionate, betamethasone 17-propionate, calcipotriol, and MC1080. Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, and no subjects had enough positive samples to allow calculation AUC(0-t) for betamethasone dipropionate. Betamethasone 17-propionate was only detected in 12 samples from 5 subjects, and only 2 subjects had enough positive samples to calculate AUC(0-t). The mean value of AUC(0-t) for these 2 subjects is presented for betamethasone 17-propionate. Calcipotriol and MC1080 were never detected above lower limit of quantification, therefore no PK parameters could be calculated and no data have been entered for calcipotriol and MC1080.
Time Frame: Week 4, blood samples taken before IMP was applied and 1, 3, and 5 hours after application of IMP
Population: PK evaluation was performed in 32 subjects. Analysis set not defined in clinical trial protocol.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 32
pg*h/mL
  Betamethasone dipropionate: number analyzed (Participants) | 4
  Betamethasone dipropionate | NA (NA) — Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, therefore it was not possible to calculate AUC(0-t).
  Betamethasone 17-propionate: number analyzed (Participants) | 5
  Betamethasone 17-propionate | 325 (193.75)

18. Secondary Outcome: Pharmacokinetic Evaluation AUC(0-infinity)
Description: AUC(0-infinity) values for betamethasone dipropionate, betamethasone 17-propionate, calcipotriol, and MC1080. Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, and no subjects had enough positive samples to allow calculation AUC(0-infinity) for betamethasone dipropionate. Betamethasone 17-propionate was only detected in 12 samples from 5 subjects, and only 2 subjects had enough positive samples to calculate AUC(0-infinity). The mean value of AUC(0-infinity) for these 2 subjects is presented for betamethasone 17-propionate. Calcipotriol and MC1080 were never detected above lower limit of quantification, therefore no PK parameters could be calculated and no data have been entered for calcipotriol and MC1080.
  The terms AUC(0-infinity) and AUC(all) are interchangeable, AUC(0-infinity) was used in the protocol whereas AUC(all) was used in the report. AUC(0-infinity) has been used here to be consistent with the protocol.
Time Frame: Week 4, blood samples taken before IMP was applied and 1, 3, and 5 hours after application of IMP
Population: PK evaluation was performed in 32 subjects. Analysis set not defined in clinical trial protocol.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 32
pg*h/mL
  Betamethasone dipropionate: number analyzed (Participants) | 4
  Betamethasone dipropionate | NA (NA) — Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, therefore it was not possible to calculate AUC(0-infinity).
  Betamethasone 17-propionate: number analyzed (Participants) | 5
  Betamethasone 17-propionate | 325 (193.75)

19. Secondary Outcome: Pharmacokinetic Evaluation C(Max)
Description: C(max) values for betamethasone dipropionate, betamethasone 17-propionate, calcipotriol, and MC1080. Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects and betamethasone 17-propionate was only detected in 12 samples from 5 subjects, therefore pharmacokinetic profiles could not be calculated. Presented C(max) values for betamethasone dipropionate and betamethasone 17-propionate are the the single highest concentrations measured in any sample at any time. Calcipotriol and MC1080 were never detected above lower limit of quantification, therefore no PK parameters could be calculated and no data have been entered for calcipotriol and MC1080.
Time Frame: Week 4, blood samples taken before IMP was applied and 1, 3, and 5 hours after application of IMP
Population: PK evaluation was performed in 32 subjects. Analysis set not defined in clinical trial protocol.
Measure: Number; unit: pg/mL
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 32
pg/mL
  Betamethasone dipropionate: number analyzed (Participants) | 4
  Betamethasone dipropionate | 104
  Betamethasone 17-propionate: number analyzed (Participants) | 5
  Betamethasone 17-propionate | 126

20. Secondary Outcome: Pharmacokinetic Evaluation T(Max)
Description: T(max) values for betamethasone dipropionate, betamethasone 17-propionate, calcipotriol, and MC1080. Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects and betamethasone 17-propionate was only detected in 12 samples from 5 subjects. Therefore it was not possible to calculate T(max) for betamethasone dipropionate and betamethasone 17-propionate. Calcipotriol and MC1080 were never detected above lower limit of quantification, therefore no PK parameters could be calculated and no data have been entered for calcipotriol and MC1080.
Time Frame: Week 4, blood samples taken before IMP was applied and 1, 3, and 5 hours after application of IMP
Population: PK evaluation was performed in 32 subjects. Analysis set not defined in clinical trial protocol.
Measure: Number; unit: h
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 32
h
  Betamethasone dipropionate: number analyzed (Participants) | 4
  Betamethasone dipropionate | NA — Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, therefore it was not possible to calculate T(max).
  Betamethasone 17-propionate: number analyzed (Participants) | 5
  Betamethasone 17-propionate | NA — Betamethasone 17-propionate was only detected above lower limit of quantification in 12 samples from 5 subjects, therefore it was not possible to calculate T(max).

21. Secondary Outcome: Pharmacokinetic Evaluation T(½)
Description: T(½) values for betamethasone dipropionate, betamethasone 17-propionate, calcipotriol, and MC1080. Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects and betamethasone 17-propionate was only detected in 12 samples from 5 subjects, therefore it was not possible to calculate T(½) for betamethasone dipropionate or betamethasone 17-propionate. Calcipotriol and MC1080 were never detected above lower limit of quantification, therefore no PK parameters could be calculated and no data have been entered for calcipotriol and MC1080.
Time Frame: Week 4, blood samples taken before IMP was applied and 1, 3, and 5 hours after application of IMP
Population: PK evaluation was performed in 32 subjects. Analysis set not defined in clinical trial protocol.
Measure: Number; unit: h
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 32
h
  Betamethasone dipropionate: number analyzed (Participants) | 4
  Betamethasone dipropionate | NA — Betamethasone dipropionate was only detected above lower limit of quantification in 5 samples from 4 subjects, therefore it was not possible to calculate T(½).
  Betamethasone 17-propionate: number analyzed (Participants) | 5
  Betamethasone 17-propionate | NA — Betamethasone 17-propionate was only detected above lower limit of quantification in 12 samples from 5 subjects, therefore it was not possible to calculate T(½).

22. Secondary Outcome: Subjects With "Controlled Disease" According to the Investigator's Global Assessment of Disease Severity on the Body at End of Treatment
Description: Subjects with "Controlled disease" (i.e., "Clear" or "Almost clear" for subjects with at least "Moderate" disease at baseline, "Clear" for subjects with "Mild" disease at baseline) according to the investigator's global assessment of disease severity on the body at end of treatment, defined as the last value recorded up to and including Week 8.
Time Frame: End of treatment
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Participants
  Controlled | 62
  Non-controlled | 45

23. Secondary Outcome: Percentage Change in PASI From Baseline to End of Treatment
Description: Percentage change in Psoriasis area and severity index (PASI) score from baseline to end of treatment, defined as the last value recorded up to and including Week 8. Psoriasis area and severity index (PASI) assesses extent and severity of clinical signs of psoriasis vulgaris. Body surface is divided in 4 ares: head (incl. neck), arms (incl. hands), trunk (incl. flexures) and legs (incl. buttocks and feet). Each area is scored from 0-6 for extent of psoriasis and from 0-4 for redness, thickness, and scaliness, and an area PASI score is calculated. The total PASI score is calculated from each area's score. The PASI score ranges from 0 (clear skin) to 72 (maximum disease), a PASI score higher than 10 generally corresponds to moderate-to-severe disease.
Time Frame: From baseline to end of treatment
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Percentage change in PASI score
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Percentage change in PASI score | -78.7 (32.4)

24. Secondary Outcome: Subjects With "Controlled Disease" According to the Patient's Global Assessment of Disease Severity on the Body at End of Treatment
Description: Subjects with "Controlled disease" (i.e., "Clear" or "Almost clear" for subjects with at least "Moderate" disease at baseline, "Clear" for subjects with "Mild" disease at baseline) according to the patient's global assessment of disease severity on the body at end of treatment, defined as the last value recorded up to and including Week 8.
Time Frame: End of treatment
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 107
Participants
  Controlled | 67
  Non-controlled | 40

ADVERSE EVENTS:
Time Frame: During the trial, the investigator followed up all AEs (SAEs) until the final outcome was determined. After a subject had left the trial, the investigator followed up all non-serious AEs classified as possibly or probably related to the IMP for 14± 2 days or until the final outcome was determined, whichever came first. SAEs were followed up until a final outcome had been determined, that is, the follow-up could continue beyond the end of the trial.
Arm/Group | LEO 80185 Gel
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 1/107
Other Adverse Events (participants affected / at risk) | 38/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 80185 Gel (N=107)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 80185 Gel (N=107)
Nasopharyngitis (Infections and infestations) | 6 (6)
Rhinitis (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Blood parathyroid hormone increased (Investigations) | 4 (5)
Blood cortisol decreased (Investigations) | 2 (2)
Eosinophil count increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 6 (8)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.

DOCUMENTS (2):
  • Study Protocol (2013-04-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT02038569/Prot_001.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT02038569/SAP_000.pdf